CLINICAL TRIAL: NCT05790525
Title: Effect of Oral Helicobacter Pylori Infection on the Efficacy of Gastroluminal Helicobacter Pylori Eradication Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Principal Investigator, Clinical Professor, Xijing Hospital of Digestive Diseases
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20232027-C-1-B
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Helicobacter Pylori
Keywords: Oral Helicobacter pylori; Helicobacter pylori gastric; Eradication rate of Helicobacter pylori in the stomach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Both gastric and oral Helicobacter pylori are positive (Other)
  Interventions: Drug: Standard bismuth quadruple
- Positive for Helicobacter pylori for gastric and negative for Helicobacter pylori for oral cavity (Other)
  Interventions: Drug: Standard bismuth quadruple

INTERVENTIONS:
Drug: Standard bismuth quadruple — Use the standard bismuth quadruple regimen recommended by the latest Chinese guidelines

SUMMARY:
The aim of this study is to assess the effect of oral Helicobacter pylori infection on the efficacy of gastric Helicobacter pylori infection eradication. Patients diagnosed with gastric Helicobacter pylori infection are tested for oral Helicobacter pylori and given standard bismuth quadruple therapy, with a urea breath test, a rapid urease test, or a Helicobacter pylori stool antigen test to confirm gastric Helicobacter pylori eradication at week 6 follow-up, and an oral Helicobacter pylori test kit to confirm oral Helicobacter pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18~70 ,both gender.
2. Initial diagnosis of stomach Helicobacter pylori infection or never had Helicobacter pylori infection.
3. Have not received dental care or systemic periodontal basic treatment in the past 1 year.

Exclusion Criteria:

1. Those who have contraindications to the drugs used in this institute or are allergic to the drugs used.
2. There is serious organ damage and complications (such as cirrhosis, uremia, etc.), severe or unstable cardiopulmonary or endocrine diseases.
3. Ongoing use of antiulcer medications (including PPIs taken within 2 weeks before Helicobacter pylori infection testing), antibiotics, or bismuth complexes (more than 3 times/week before screening).
4. Those with severe oral diseases and malignant tumors of the mouth.
5. Women planning pregnancy, pregnancy and breastfeeding.
6. Previously had upper gastrointestinal surgery.
7. Those who do not take their medication on time.
8. Refusal to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori in the stomach | 28 days after treatment
  The primary end point of this study is to compare the rate of gastric Helicobacter pylori eradication in oral Helicobacter pylori positive and negative

SECONDARY OUTCOMES:
Oral Helicobacter pylori conversion rate | 28 days after treatment
  Oral Helicobacter pylori conversion rate 28 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Shi, PhD, Study Director — Xijing Hosipital of Digestive Disease
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China